CLINICAL TRIAL: NCT04108481
Title: Immunotherapy Combined With Yttrium-90 RadioEmbolization in the Treatment of Colorectal Cancer With Liver Metastases [iRE-C - Clinical Trial]
Brief Title: Immunotherapy With Y90-RadioEmbolization for Metastatic Colorectal Cancer
Acronym: iRE-C
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: DSMC-directed closure
Sponsor: University of Iowa (Other)
Collaborators: Biocompatibles UK Ltd (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201909709
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer Metastatic; Colon Cancer; Metastatic Colorectal Cancer; Rectal Cancer; Liver Metastasis Colon Cancer; Colo-rectal Cancer; Colorectal Adenocarcinoma; Colorectal Neoplasms; Liver Metastases; Colorectal Carcinoma
Keywords: Y90; Y90-RE; Radioembolization; Y90-Radioembolization; y-90; Yttrium; Yttrium-90; Microsatellite Stable; MSS; CRC; mCRC; Colorectal; Liver Metastases; Liver Metastasis; Durvalumab; Anti-PD1; Anti-PDL1; Immunotherapy; Colorectal Cancer; Mismatch repair proficient; pMMR; KRAS; NRAS; BRAF; BRAF-V600E
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms | interventions — durvalumab; atezolizumab; Yttrium-90

STUDY DESIGN:
Intervention Model Description: Accelerated titration design with an expansion phase once MTD is determined to treat up to a total of 18 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Y90-RE in combination with immunotherapy (durvalumab) (Experimental): The treatment phase starts of with the immunotherapy drug (durvalumab) - "priming doses" every 2 weeks prior to patient getting mapped and ready for treatment with Y90-RadioEmbolization.
  Post-Y90-RE, treatment is approximately 2 months in combination with fixed doses (750 mg) of durvalumab. The number and timing of doses of durvalumab each patient will receive will depend on the dose level the patient is assigned to (range 2-5 doses of immunotherapy).
  A single patient will be treated per dose level until the first dose limiting toxicity (DLT) is recorded. Once the first DLT is recorded, two additional patients are treated at the same dose level and the trial reverts to a standard 3+3 design. Up to 6 patients will be treated at each dose level. The maximum tolerated dose (MTD) will be defined as the highest dose level for which at most 1 out of 6 patients experience a DLT.
  Interventions: Drug: Durvalumab; Radiation: Yttrium-90 RadioEmbolization

INTERVENTIONS:
Drug: Durvalumab — Immunotherapy
  Other Names: IMFINZI; MEDI4736; MEDI-4736; Anti-PDL1
Radiation: Yttrium-90 RadioEmbolization — Microscopic radioactive particles (TheraSphere®) will be used for radioembolization to deliver the Y90 drug to the liver
  Other Names: Y90-RE; Y90; Glass Microspheres; yttrium90; Y-90 Glass Microspheres

SUMMARY:
This clinical trial will be conducted as a single-center, open-label, Phase I/2 trial to evaluate the feasibility and safety of Yttrium-90 radioembolization (Y90-RE) in combination with a fixed dose of of immunotherapy (durvalumab - 750 mg) in subjects with liver-predominant, metastatic colorectal cancer (mCRC), which is mismatch repair proficient/microsatellite stable (pMMR/MSS).

DETAILED DESCRIPTION:
The purpose of this clinical trial is to find out more about the side effects of immunotherapy with a form of radiation treatment for the cancer in the liver called Yttrium-90 RadioEmbolization (Y90-RE). An immunotherapy drug, durvalumab, will be given intravenously every 2 weeks. Investigators are studying what doses of durvalumab are safe for people in combination with this form of radiation treatment. Patients in this study will receive durvalumab, which is experimental and not approved by the U.S. Food and Drug Administration (FDA) for metastatic colorectal cancer. Microscopic radioactive particles (TheraSphere®) will be used for radioembolization to deliver the Y90 drug to the liver.

The number of doses of the immunotherapy drug (range: 2 to 5) will depend on the cohort patients are assigned to. There is no placebo. Everyone on the study is treated with immunotherapy alongside Y90-RadioEmbolization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histological or cytological confirmation of colorectal cancer with metastasis to the liver. Mismatch repair or microsatellite instability status of the tumor needs to be known. Tumors need to be mismatch repair proficient (for mismatch repair deficient tumors immunotherapy is already approved).
* Patient must have at least 1 liver lesion measurable as defined in the protocol
* Must have liver metastases and be appropriate for treatment with Y-90 radioembolization therapy as determined by the treating medical oncologist and interventional radiologist/oncologist, and nuclear medicine physician(s). NOTE: the goal of therapy is safety and parenchymal sparing. Typically, since the treatment is personalized, the goal is to have at least 30% liver parenchymal sparing post treatment.
* Must have a metastatic focus amendable to biopsy. It is permissible to use same or alternative lesion for biopsy for assessment for tumor response and changes in microenvironment (mandatory pre- and post-Y90-RE biopsy).
* At least 2 but no more than 3 lines of therapy allowed in metastatic setting. These include at least treatment with a fluoropyrimidine, oxaliplatin, and/or irinotecan-based therapy, an anti-VEGF therapy and, if RAS wild-type, an anti-EGFR therapy, unless deemed intolerant or not suitable by the treating oncologist. NOTE: adjuvant and/or maintenance chemotherapy does not count as an additional line of therapy. (Patients with more than 3 lines of therapy are at risk for liver disease from prior systemic therapies and would not be reasonable candidates for Y90-RE).
* ECOG Performance Status (PS) 0 or 1.
* Negative serum pregnancy test done ≤7 days prior to registration, for persons of childbearing potential only.
* Females of childbearing potential (FOCBP), must use appropriate method(s) of contraception. FOCBP are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause). Additionally, FOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with durvalumab plus 5 half-lives of durvalumab (13 weeks) plus 30 days (duration of ovulatory cycle) for a total of 17 weeks post-treatment completion (details in appendix).
* Men who are sexually active with FOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with durvalumab plus 5 half-lives of durvalumab plus 90 days (duration of sperm turnover) for a total of 25 weeks post-treatment completion (details in appendix).
* Provide written informed consent.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Willingness to provide mandatory blood specimens for correlative research (detailed in protocol).
* Willingness to provide mandatory tissue specimens for correlative research (detailed in protocol). NOTE: If tissue is deemed inaccessible, patient cannot participate in study.
* Willingness to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
* Must have a life expectancy of at least 6 months.

Exclusion Criteria:

* Any of the following laboratory abnormalities:

  * Hemoglobin <8.0 g/dL
  * Absolute neutrophil count (ANC) <1500/mm3
  * Platelet count <100,000/mm3
  * Total bilirubin >1.5 x ULN (except in subjects with Gilbert Syndrome, who cannot have a total bilirubin > 3.0 mg/dL)
  * Alanine aminotransferase (ALT) and Aspartate transaminase (AST) >2.5 x ULN
  * Serum creatinine > 1.5 x ULN OR
  * Calculated creatinine clearance <30 ml/min using the Cockcroft-Gault formula
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic infections, or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Untreated central nervous system (CNS) metastatic disease (including spinal cord and leptomeningeal disease). NOTE: Patients with previously treated CNS metastases that are radiographically and neurologically stable for ≥ 6 weeks are permitted.
* Uncontrolled intercurrent illness including, but not limited to, autoimmune disease, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements. EXCEPTION: Patients who have adequately controlled autoimmune disease with or without medications are permitted as long as deemed reasonable by treating physician.
* Received any other investigational agent incorporating chemotherapy and/or biologics within 14 days prior to first dose of durvalumab which would be considered as a treatment for the primary neoplasm. For patients on active treatment, last treatment and 1st dose of Durvalumab should be at least ≥ 14 days. EXCEPTION: Other forms of concurrent observational studies are permitted.
* Other active malignancy ≤3 years prior to registration. EXCEPTIONS: Non-melanoma skin cancer, lentigo maligna- in-situ, or carcinoma-in-situ of the cervix. Also prior malignancy already treated with curative intent and with no known active disease present would be considered eligible.
* History of unstable cardiac disease defined as one of the following:

  * Congestive heart failure > class II New York Heart Association (NYHA). (Appendix II)
  * Unstable angina (angina symptoms at rest) or new onset angina (began ≤ 3 months prior to registration)
  * Myocardial infarction ≤ 3 months
  * Uncontrolled cardiac ventricular arrhythmias. EXCEPTION: Subjects that are stable on anti-arrhythmic therapy are eligible.
* Any concurrent chemotherapy, biologic, or hormonal therapy for cancer treatment within 14 days of first dose of durvalumab. NOTE: Subjects can be screened during washout period.
* History of severe allergic reactions (i.e. Grade 4 allergy, anaphylactic reaction from which the subject did not recover ≤ 6 hours of initiation of supportive care)
* Failure to recover from toxicities from prior anti-cancer therapy, defined as having not resolved to National Cancer Institute (NCI) CTCAE version 5.0 Grade ≤ 1. EXCEPTIONS: Alopecia and laboratory values listed per the exclusion criteria. Also subjects with irreversible toxicity that is not reasonably expected to be exacerbated by any investigational products (i.e. hearing loss) will be permitted.
* Use of steroids. EXCEPTIONS: Systemic glucocorticoids will be permitted as long as it is ≤20 mg of prednisone equivalent. Topical steroids, such as bronchodilators and local steroid injections are also permitted if clinically required.
* Patients with renal failure currently requiring dialysis of any kind.
* Patients weighing <30kg will be excluded from enrollment
* History of allogenic organ transplantation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of Yttrium-90 radioembolization combined with immunotherapy durvalumab to treat liver-predominant metastatic colorectal cancer (mCRC) | Initiation of treatment up to 8 weeks and 2 doses ("priming") of immunotherapy prior to Y90-RE.
  MTD will be defined as the highest dose level for which at most 1 out of 6 patients experience a dose-limiting toxicity (DLT) using CTCAE version 5.0.

SECONDARY OUTCOMES:
Incidence of adverse events (AE) per CTCAE version 5.0 | Initiation of screening up to 2 years
  The number and severity of all adverse events (overall, by dose-level, and by tumor molecular subtype) will be tabulated and summarized.
Determine overall response rate (ORR) | Up to 2 months post treatment
  Overall response rate is defined as the proportion of evaluable patients that have achieved a complete response (CR) or partial response (PR) by RECIST v1.1 as well as mRECIST and iRECIST.
Determine the disease control rate (DCR) | Up to 2 months post treatment
  Disease control rate is defined as the proportion of evaluable patients that have achieved a complete response (CR), partial response (PR), or stable disease (SD) by RECIST v1.1 as well as mRECIST and iRECIST.
Determine liver-specific progression free survival | Up to 2 months post treatment
  Progression free survival is defined as the proportion of evaluable patients that have achieved liver-specific progression free survival (Liver-PFS)
Determine overall progression free survival | Up to 2 years
  Progression free survival is defined as the proportion of evaluable patients that have achieved overall progression free survival (PFS)
Determine overall survival | Up to 2 years
  Overall survival (OS) is defined as the time from randomization to death of any cause.
Determine duration of response | Up to 2 years
  Duration of response (DOR) is defined as the time measurement criteria for CR or PR (whichever status is recorded first) until the first date that recurrence or PD is objectively documented, taking as reference for PD the smallest measurements recorded since the treatment started.

OTHER OUTCOMES:
Circulating tumor DNA - ctDNA - liquid biopsy correlates | Up to 2 months post treatment
  To determine changes in the expression profile and in levels of circulating tumor DNA (ctDNA) in blood pre- and post- treatment
Immune correlates - tissue | Up to 2 months post treatment
  To assess the changes in immune infiltration (TISSUE: tumor-infiltrating lymphocytes - TILs (CD-3, CD-8), PD-L1 and PD-1 expression, pre- and post-Y90-RE and immunotherapy)
Immune correlates - blood | Up to 2 months post treatment
  To analyze serial changes in immune cells (BLOOD) pre- and post-Y90-RE and immunotherapy
Tumor tissue - correlates | Up to 2 months post treatment
  To evaluate mutation burden by whole-exome sequencing pre- and post-treatment (TISSUE)
Tumor tissue - correlates | Up to 2 months post treatment
  To evaluate concomitant expression profile changes through RNA-Seq pre- and post-treatment (TISSUE)
Abscopal effects | Up to 2 months post treatment
  To report on any abscopal effects seen in terms of responses outside the Y90-RE field

CONTACTS AND LOCATIONS:
Overall Officials: Chandrikha Chandrasekharan, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT04108481/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT04108481/ICF_001.pdf